CLINICAL TRIAL: NCT02539901
Title: Cognitive and Communicative Development Description of Deaf Child With a Cochlear Implant.
Brief Title: Development of a Deaf Child With a Cochlear Implant.
Acronym: DECCODES
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 11 227 02; 2011-A01058-33 (Registry Identifier: Agence National du Médicament et des Produits de santé)
Record Dates: First submitted 2015-08-18; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Deafness
Keywords: cochlear implant; Developmental Psychology; cognitive development; communicative development; perceptual development; deaf child
MeSH Terms: conditions — Deafness | interventions — Neuropsychological Tests; Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 12-30 months-old deaf children: Children with deafness of bilateral deep perception had : Evaluation of the detection of non-linguistic sounds, Early Social Communication Scale (ECSP) and psychomotor infancy development scale or Lézine Brunet-Revised scale
  Interventions: Behavioral: Evaluation of the detection of non-linguistic sounds; Behavioral: Early Social Communication Scale (ECSP); Behavioral: psychomotor infancy development scale
- 6-9 years-old deaf children: Free hearing test categorization and NEPSY (two domains: "memory and learning" and "attention and executive functions") in 6-9 years-old deaf child cohort with deafness of bilateral deep perception and carrying a cochlear implant
  Interventions: Behavioral: Free hearing test categorization; Behavioral: NEPSY (two domains: "memory and learning" and "attention and executive functions").
- 12-30 months-old normal hearing children: Evaluation of the detection of non-linguistic sounds in 12-30 months-old normal hearing child cohort
  Interventions: Behavioral: Evaluation of the detection of non-linguistic sounds
- 6-9 years-old normal hearing children: 'Free hearing test categorization' in 6-9 years-old normal hearing child cohort
  Interventions: Behavioral: Free hearing test categorization

INTERVENTIONS:
Behavioral: Evaluation of the detection of non-linguistic sounds — Evaluation of the detection of non-linguistic sounds (sound room)
  Groups: 12-30 months-old deaf children; 12-30 months-old normal hearing children
Behavioral: Free hearing test categorization — Free hearing test categorization evaluation
  Groups: 6-9 years-old deaf children; 6-9 years-old normal hearing children
Behavioral: Early Social Communication Scale (ECSP) — Early Social Communication Scale (ECSP) evaluation
  Groups: 12-30 months-old deaf children
Behavioral: psychomotor infancy development scale
  Other Names: Lézine Brunet-Revised scale
  Groups: 12-30 months-old deaf children
Behavioral: NEPSY (two domains: "memory and learning" and "attention and executive functions"). — NEPSY evaluation
  Groups: 6-9 years-old deaf children

SUMMARY:
Cochlear implantation enables profoundly deaf children to acquire speech and develop their understanding of spoken language. However, there are significant interindividual differences in the results obtained with the implant. Given the lack of theoretical knowledge on acoustic predictors, cognitive and language to obtain optimum speech recognition with cochlear implants associated with a good communicative and language development of deaf children, the investigators intend to achieve a preliminary longitudinal study aimed to describe the cognitive, communicative and perceptive implanted deaf children.

The main objective of our study is to describe the cognitive and communicative development of deaf children implanted from the pre-implant assessment to 18 months post-implantation, by addressing the following aspects:

* The psychomotor and cognitive development assessed using the Brunet-Lézine test;
* The development of preverbal communication, evaluated using the Early Social Communication Scale.

ELIGIBILITY:
INCLUSION CRITERIA:

To achieve this study, two cohorts will be formed:

* A cohort of deaf children aged 12 to 30 months:

  * Be reached a bilateral profound sensorineural hearing loss (greater than 90 dB hearing loss, as classified by the International Bureau for Audiophonology, 1997);
  * Raise a cochlear implant;
  * Being affiliated to a social security scheme.
  * Consent representatives of parental authority (or at least one of the two)
* A cohort of deaf children from 6 to 9 years:

  * Be reached a bilateral profound sensorineural hearing loss;
  * Be holder of a cochlear implant for at least 3 years;
  * Consent representatives of parental authority (or at least one of the two).
* A group of normal hearing typically developing children:

this group will provide benchmarks for perception tests. It consists of two sub-groups:

* Children with normal hearing typically developing 12 to 30 months; children whith a general, linguistic and normal psychomotor evaluated on the basis of prior clinical examination at baseline and on the compilation of their health record. They must not present psychomotor retardation or language.
* Children with normal hearing in typical development 6 to 9 years.

  * Be matched in age and sex with deaf children (a pairing with a child on the criteria defined above). In terms of developmental age, we can consider as having comparable in terms of age development of children with:
  * +/- 6 months for the population of children 6 to 9 years
  * +/- 1 month for the population of children 12 to 30 months.
  * Have a typical development, evaluated by a grade level for their age;
  * Consent representatives of parental authority (or at least one of the two).

EXCLUSION CRITERIA:

Will be excluded from our study subjects where there is an inability to meet the tests, either in situations:

* Impossible to understand instructions
* Blindness
* Impossible to meet the tests
* Multihandicap
* A legal impossibility. Furthermore, children will be excluded for which there is a refusal on the part of the parents or of the child to participate in the study (for children old enough to express their opinion).

Ages: 12 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Young patients consulting in the Unit of Pediatric Cochlear Implantation, Hospital-University Centre of Toulouse.
  The normal hearing participants will be recruited by posters, produced in various places childcare (crèches, schools) or pediatric services Purpan hospital.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
screening and diagnosis of global developmental delays in young children | inclusion
evaluation of variation pre-linguistic communication and lexicon emergence | inclusion, 6 months, 12 months and 18 months

SECONDARY OUTCOMES:
Non-linguistic variation of sounds Detection Test | inclusion, 6 months, 12 months and 18 months
Neuropsychological assessment of child development variation | inclusion, 6 months, 12 months and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DEGUINE, MD, PhD, Principal Investigator — Service ORL - Hôpital Purpan
Locations (1):
- Hôpital Purpan - Pavillon Dieulafoy - Service ORL (ENT services), Toulouse, Haute-Garonne, France